CLINICAL TRIAL: NCT05544539
Title: the Effect of Ozone Oil on the Post Operative Sequelae After Surgical Removal of Impacted Mandibular Third Molar: Randomized Clinical Trial
Brief Title: the Effect of Ozone Oil on the Postoperative Sequalae After Surgical Removal of Third Molar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Maiyada A. Talib, dentist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mandibular third molar
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Impacted Third Molar Tooth
Keywords: third molar; ozone oil
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug arm (Experimental): In the study group the (0.5 ml) of Ozone oil (perio3®, Hoffmann, German) was placed inside the socket of the extracted tooth filling it completely following suturing of the flap
  Interventions: Drug: Ozone-Based Agent
- placebo arm (Placebo Comparator): the ozone oil syringe was placed inside the patient mouth without applying the oil.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ozone-Based Agent — In the study group Ozone oil was placed inside the socket of the extracted tooth following suturing of the flap
  Other Names: ozone
  Arms: drug arm
Drug: Placebo — In the control group Ozone oil syringe was placed inside the socket of the extracted tooth without applying the oil
  Arms: placebo arm

SUMMARY:
This study aimed to evaluate the effectiveness of intra socket application of Ozone oil on postoperative pain, trismus and facial swelling following the surgical extraction of impacted mandibular third molars.

DETAILED DESCRIPTION:
Background: Surgical removal of impacted teeth is frequently encountered in dental clinic. Pain, trismus, and swelling are common postoperative sequelae for third molar surgery. Different methods have been used to prevent or decrease these postoperative sequelae, one of them is the application of Ozone oil that shows many advantages in controlling the inflammation, thus reducing pain, trismus and swelling. There is an evidence to suggest that it may have significant effects in the synthesis, release, and metabolism of a series of biochemical substances.

Aim of the study: This study aimed to evaluate the effects of local application of Ozone oil on postoperative pain, trismus and facial swelling following the surgical removal of mandibular third molars.

Materials and Methods: This triple blind randomized prospective clinical trial was performed during period from January 2021 until the end of July 2021, on (40) patients, age range was between (18-35) years, with impacted mandibular third molar in similar positions (Class I-II and position B, Pell and Gregory's classification). They were randomly assigned into two groups, 20 patients for Ozone oil group treated with topical application of Ozone oil in their socket, and 20 patients into the control group in which the Ozone oil syringe was inserted inside the patient mouth without applying the treatment. Assessment of trismus was done by measuring the maximum mouth opening and the swelling was assessed by measuring distance between five predetermined points (tragus, angle of mouth, pogonion, lateral angle of eye and angle of mandible). These measurements were done before surgery as a baseline record as well as at the second and seventh postoperative days. Pain was evaluated using numeric rating scale from the day of surgery until the seventh day.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with mandibular third molar (Class I-II and position B, Pell and Gregory's classification) 2. Patients who were willing to compliance with study 3. the Surgical site free of active infection. 4. patients without any systemic disease that might affect the healing process such as uncontrolled diabetes.

Exclusion Criteria:

* 1. Medical condition that prevent surgical intervention such as patient with bleeding disorders, recent myocardial infarction, psychiatric problem, uncontrolled systemic diseases, and patients with pacemaker, immunocompromised status and who were taking corticosteroidand anti-inflammatory drugs.

  2.. Poor oral hygiene and/or active advanced periodontal disease and, or patients with active local infection in relation to the third molar such as Pericoronitis.

  3. Smokers. 9. Any systemic condition that interfere with the use of ozone such as autoimmune disorders, myasthenia, hyperthyroidism, myocardial infarction, alcohol intoxication and ozone allergy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
measuring pain severity after extraction using numerical rating scale | 7 days
  severity measured using numerical rating scale from the first postoperative day to 7th day
assessing the change in mouth opening using vernier caliper | baseline , the 2nd and 7th postoperative day
  severity, baseline , the 2nd and 7th postoperative day
measuring the change in facial measurement to assess the swelling | baseline , the 2nd and 7th postoperative day
  severity, baseline , the 2nd and 7th postoperative day

SECONDARY OUTCOMES:
surgical difficulty | through out the operation duration, an average of 1 hour
  duration and technique
class | through out the operation duration, an average of 1 hour
  cl 1 and cl 2
angulation of impaction | through out the operation duration, an average of 1 hour
  mesioangular , vertical, horizontal

CONTACTS AND LOCATIONS:
Overall Officials: Maiyada Talib, Principal Investigator — Baghdad university
Locations (1):
- Baghdad University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No